CLINICAL TRIAL: NCT02706067
Title: Multifactorial Approach Associated With Orlistat (Xenical) for 4 Years Weight Loss Maintenance in Obese Patients
Brief Title: Multifactorial Approach Associated With Orlistat (Xenical) for 4 Years Weight Loss Maintenance in Obese Adults
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML16868
Record Dates: First submitted 2016-03-08; First posted 2016-03-11 (Estimated); Last update posted 2016-04-05 (Estimated); Status verified 2016-04

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Orlistat

ARMS (1):
- Orlistat (Experimental): Participants will receive intermittent orlistat for up to 4 years, with the dose determined according to body weight changes.
  Interventions: Drug: Orlistat

INTERVENTIONS:
Drug: Orlistat — Participants will receive orlistat on an intermittent basis as 120 milligrams (mg) three times a day: once with breakfast, once with lunch, and once with dinner. In case of weight relapse (increase 2.5 percent [%] or more from Baseline) orlistat will be administered for up to 2 months or until weight regain reaches 0% from Baseline. For special occasions (feasts, birthdays, anniversaries) orlistat will be given for up to 3 days.
  Other Names: Xenical

SUMMARY:
This study will evaluate the efficacy of a multifactorial approach associated with orlistat (Xenical) in weight loss maintenance during 4 years. The effect of orlistat in combination with diet, physical activity, and/or cognitive behavioral therapy will be monitored.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) greater than or equal to (>/=) 30 kilograms per meter-squared (kg/m^2), or BMI >/= 28 kg/m^2 with risk factors of diabetes, hypertension, or hyperlipidemia, before weight loss
* Documented weight loss >/= 10% of initial body weight obtained with diet, with or without psychological therapy or orlistat

Exclusion Criteria:

* Pregnant or lactating females
* History or presence of significant medical disorders
* Active gastrointestinal disorders such as peptic ulcer disease or malabsorption syndromes
* Pancreatic disease: pancreatic enzyme deficiency, history or current presence of pancreatitis
* Clinically significant abnormal clinical chemistry or hematology results
* Excessive alcohol intake
* Smoking cessation within the previous 6 months
* History or presence of cancer
* Administration of medicines known to alter body weight
* History or presence of cancer

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2002-07; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Percent Change from Baseline in Body Weight at Year 2 | Baseline and Year 2
Percent Change from Baseline in Body Weight at Year 4 | Baseline and Year 4

SECONDARY OUTCOMES:
Percentage of Participants Diagnosed with Binge Eating Disorder According to Diagnostic and Statistical Manual of Mental Disorders (DSM) IV Criteria | Every 6 months during Year 1, annually during Years 2 to 4
Eating Disorder Inventory (EDI) 2 Subscale and Total Score | Baseline and Year 4
Hospital Anxiety and Depression (HAD) Subscale Score | Baseline and Year 4
Number of Orlistat Capsules Taken During the Study | Given up to three times per day for 4 years
Duration of Orlistat Treatment During the Study | Given up to three times per day for 4 years
Waist-to-Hip Circumference Ratio | Baseline and Year 4
Waist, Hip, Wrist, and Arm Circumference (Expressed in Centimeters) | Baseline and Year 4
Skinfold Thickness (Expressed in Millimeters) | Baseline and Year 4
Bioelectrical Impedance (Expressed in Kilograms of Body Fat Mass) | Baseline and Year 4
Number of Kilocalories Expended, Total and at Rest | Baseline and Year 4

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Chair — Hoffmann-La Roche
Locations (1):
- Geneva, Switzerland